CLINICAL TRIAL: NCT00968422
Title: A Study of Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ABT-384 in Elderly Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Gerard Marek, MD, PhD, Abbott
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M10-506
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Last update posted 2010-11-03 (Estimated); Status verified 2010-09

CONDITIONS: Healthy
Keywords: Pharmacology; Drug Safety; Phase 1 Clinical Trials; Pharmacokinetics
MeSH Terms: interventions — N-(5-(aminocarbonyl)tricyclo(3.3.1.13,7)dec-2-yl)-alpha,alpha-dimethyl-4-(5-(trifluoromethyl)-2-pyridinyl)-1-piperazineacetamide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Low dose ABT-384 (Experimental)
  Interventions: Drug: ABT-384
- Mid dose ABT-384 (Experimental)
  Interventions: Drug: ABT-384
- High dose ABT-384 (Experimental)
  Interventions: Drug: ABT-384
- Placebo (Placebo Comparator)
  Interventions: Drug: Matching placebo to ABT-384

INTERVENTIONS:
Drug: ABT-384 — 3 escalating doses will be administered daily for 21 days
  Arms: High dose ABT-384; Low dose ABT-384; Mid dose ABT-384
Drug: Matching placebo to ABT-384 — Doses will be administered daily for 21 days
  Arms: Placebo

SUMMARY:
The objectives of this study are to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of ABT-384 in elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age is 65 years or greater
2. Judged to be in a condition of general good health based on the results of medical history, physical examination, vital signs, laboratory profile and a 12-lead ECG

Exclusion Criteria:

1. Use of protocol-prohibited medications within 2 weeks prior to study drug administration.
2. Positive urine drug screen for non-prescribed drugs of abuse including alcohol.
3. Receipt of any drug depot by injection within 30 days prior to study drug administration.
4. Receipt of any investigational product within 6 weeks prior to study drug administration.
5. History of significant sensitivity or allergy to any drug.
6. History of drug or alcohol abuse within 2 years.
7. Positive test result for HBV, HCV or HIV.
8. Estimated creatinine clearance < 30 mL/min.
9. Donation or loss of 5 mL/kg or more blood volume or receipt of any blood product within 8 weeks prior to study drug administration.
10. Current enrollment in another clinical study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-08; Primary Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability Assessments (i.e., ECG, clinical laboratory tests, vital signs, weight, AE assessment, physical and brief neurological examinations) | Days -2 through 84
Assess Pharmacokinetics (i.e., ABT-384 and possible metabolite levels) and Pharmacodynamics (i.e., biomarkers of drug effect) | Days -1 through 27

CONTACTS AND LOCATIONS:
Locations (1):
- Site Reference ID/Investigator# 23024, Orlando, Florida, United States